CLINICAL TRIAL: NCT02579538
Title: Cognitive Predictors of Persistent Post-surgical Pain (PPSP)
Brief Title: Flexibility of Cognition And Persistent Pain
Acronym: FlexCAPP
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201508145
Record Dates: First submitted 2015-09-09; First posted 2015-10-19 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
Keywords: Total Knee Arthroplasty; Thoracotomy; Mastectomy; Video-Assisted Thoracoscopic Surgery (VATS); Persistent Pain; Cognitive Flexibility
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Total Knee Arthroplasty: Patients undergoing unilateral total knee arthroplasty
- Thoracic/Breast Surgery: Patients undergoing mastectomy, thoracotomy, or video-assisted thoracoscopic surgery (VATS)

SUMMARY:
This observational study aims to determine the association between preoperative cognitive flexibility and the risk of developing PPSP by preoperative administration of cognitive tests.

DETAILED DESCRIPTION:
Postoperative pain is a normal, physiologic, protective response to tissue injury that routinely resolves after healing of the surgical site. However, in some patients, pain persists long after surgery. PPSP is a diagnosis of exclusion that has most consistently been defined as pain that (1) developed after a surgical procedure, (2) is not residual from a preexisting condition, (3) has lasted for at least two months, and (4) is not attributable to other causes. One suggested risk factor for PPSP is poorer performance on tests of cognitive flexibility. Two common tests of cognitive flexibility are the Trail Making Tests (TMT) A and B and the Color Word Matching Stroop Test (CWMST).

Three hundred patients undergoing either total knee arthroplasty or thoracotomy/mastectomy will be enrolled. During preoperative evaluation, participants will complete the TMT and CWMST. Subjects will be followed prospectively and will complete surveys at one month, six months, and one year postoperatively to assess PPSP prevalence and intensity.

ELIGIBILITY:
Total Knee Arthroplasty (TKA) patients

- Inclusion criteria: Adults age 18 to 85 undergoing unilateral TKA for osteoarthritis English as primary language

- Exclusion criteria: Bilateral procedure Unable to complete cognitive testing Surgical indication for condition other than osteoarthritis (i.e. rheumatoid arthritis, spondylarthropathy) Prior knee surgery

_________________________________________________

Thoracotomy/mastectomy patients

- Inclusion criteria: Females age 18 to 85 undergoing mastectomy for breast cancer OR Adults age 18 to 85 undergoing unilateral open thoracotomy or video-assisted thoracoscopic surgery (VATS) for any non-cardiac etiology English as primary language

- Exclusion criteria: Bilateral procedure Unable to complete cognitive testing Plan for breast reconstruction Prior breast/thoracic surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 to 85 years of age undergoing unilateral TKA for osteoarthritis, unilateral mastectomy for breast cancer, or thoracotomy or video-assisted thoracoscopic surgery for any non-cardiac indication will be recruited for participation in the study during their initial preoperative visit at the Washington University Center for Perioperative Assessment and Planning (CPAP). Patient eligibility will not be affected by the anesthetic plan including the potential use of regional anesthesia techniques.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
PPSP prevalence in relation to baseline TMT B minus A time | Six months
  The time to complete TMT B test minus the time to complete TMT A test (B-A) at baseline between patients with persistent post surgical pain at six months follow-up, compared to patients without persistent post surgical pain.
PPSP prevalence in relation to baseline Stroop interference effect test score | Six months
  The Stroop interference effect time (time to complete mixed color wording - time to complete same color wording) at baseline between patients with persistent post surgical pain at six months follow-up, compared to patients without persistent post surgical pain.

SECONDARY OUTCOMES:
Comparison of cognitive test scores and severity of PPSP between patients undergoing total knee arthroplasty vs. patients undergoing thoracotomy/mastectomy | up to one year
  Association between baseline TMT B score and Stroop color interference effect results and severity of PPSP at six months follow-up in patients undergoing total knee arthroplasty vs. patients undergoing thoracotomy/mastectomy
Multiple regression analysis | up to one year
  Association of the following risk factors with PPSP at six months: cognitive flexibility (TMT and CWMST), age, gender, BMI, type of surgery, use of regional anesthesia, presence of preoperative pain, preoperative anxiety or depression, presence of prior stressful life events, and presence of severe acute postoperative pain)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Attal N, Masselin-Dubois A, Martinez V, Jayr C, Albi A, Fermanian J, Bouhassira D, Baudic S. Does cognitive functioning predict chronic pain? Results from a prospective surgical cohort. Brain. 2014 Mar;137(Pt 3):904-17. doi: 10.1093/brain/awt354. Epub 2014 Jan 17. PMID 24441173
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Solberg Nes L, Roach AR, Segerstrom SC. Executive functions, self-regulation, and chronic pain: a review. Ann Behav Med. 2009 Apr;37(2):173-83. doi: 10.1007/s12160-009-9096-5. Epub 2009 Apr 9. PMID 19357933
- [Background] Bonanno GA, Papa A, Lalande K, Westphal M, Coifman K. The importance of being flexible: the ability to both enhance and suppress emotional expression predicts long-term adjustment. Psychol Sci. 2004 Jul;15(7):482-7. doi: 10.1111/j.0956-7976.2004.00705.x. PMID 15200633
- [Background] McCracken LM, Vowles KE. Psychological flexibility and traditional pain management strategies in relation to patient functioning with chronic pain: an examination of a revised instrument. J Pain. 2007 Sep;8(9):700-7. doi: 10.1016/j.jpain.2007.04.008. Epub 2007 Jul 5. PMID 17611162
- [Background] Wicksell RK, Olsson GL, Hayes SC. Psychological flexibility as a mediator of improvement in Acceptance and Commitment Therapy for patients with chronic pain following whiplash. Eur J Pain. 2010 Nov;14(10):1059.e1-1059.e11. doi: 10.1016/j.ejpain.2010.05.001. Epub 2010 Jun 9. PMID 20538493
- [Derived] Vila MR, Todorovic MS, Tang C, Fisher M, Steinberg A, Field B, Bottros MM, Avidan MS, Haroutounian S. Cognitive flexibility and persistent post-surgical pain: the FLEXCAPP prospective observational study. Br J Anaesth. 2020 May;124(5):614-622. doi: 10.1016/j.bja.2020.02.002. Epub 2020 Mar 10. PMID 32169255